CLINICAL TRIAL: NCT07001449
Title: Effectiveness of the 'Algo(S)Therapy' Pain Neuroscience Education Program Emphasizing Physiotherapists' Communication Skills in Patients With Chronic Musculoskeletal Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Communication-Focused Pain Neuroscience Education in Chronic Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, PhD Candidate, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10841/25
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Musculoskeletal Pain
Keywords: Pain neuroscience education; Communication skills; Chronic musculoskeletal pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNE + Communication Skills (Experimental): Participants in this group will receive an individualized Pain Neuroscience Education (PNE) program plus usual physiotherapy care delivered by physiotherapists who completed the full "Algo(S)Therapy" training. This training included education in the neurophysiology of pain, assessment and management of chronic musculoskeletal pain, as well as the development and application of communication skills. The communication training focused on strategies such as motivational interviewing, empathy, active listening, and patient-centered interaction specifically tailored for individuals with chronic pain. The intervention will be administered over a 5-week period, with 2 sessions per week.
  Interventions: Behavioral: Pain Neuroscience Education with Communication Training
- PNE without Communication Training (Experimental): Participants in this group will receive an individualized Pain Neuroscience Education (PNE) intervention plus usual physiotherapy care, delivered by physiotherapists who completed only the pain neurophysiology and clinical management components of the "Algo(S)Therapy" program. These physiotherapists did not receive any formal training in communication skills, such as motivational interviewing or empathy techniques. The intervention will be administered over a 5-week period, with 2 sessions per week.
  Interventions: Behavioral: Pain Neuroscience Education without Communication Training
- Usual Physiotherapy Treatment (Active Comparator): Participants in this group will receive usual physiotherapy care. Physiotherapists in this group have not received any training in Pain Neuroscience Education or communication techniques related to chronic pain management. No components of the "Algo(S)Therapy" program will be applied in this group.
  Interventions: Behavioral: Usual Physiotherapy Treatment

INTERVENTIONS:
Behavioral: Pain Neuroscience Education with Communication Training — This intervention includes individualized physiotherapy based on a Pain Neuroscience Education (PNE) framework delivered by physiotherapists who completed the full "Algo(S)Therapy" training program. The training includes education in the neurophysiology of pain, clinical reasoning for chronic musculoskeletal pain management, and structured communication skills development (e.g., motivational interviewing, empathy, active listening). The intervention is delivered twice per week over 5 weeks (10 sessions total).
  Arms: PNE + Communication Skills
Behavioral: Pain Neuroscience Education without Communication Training — A structured PNE program focusing on the neurophysiology and clinical management of chronic musculoskeletal pain. Delivered by physiotherapists trained only in the scientific modules of the "Algo(S)Therapy" program. Does not include communication skills training. Includes 10 sessions (2/week for 5 weeks), alongside standard physiotherapy care.
  Arms: PNE without Communication Training
Behavioral: Usual Physiotherapy Treatment — Usual care based on medical referral and physiotherapy assessment. Delivered by physiotherapists who have not received training in Pain Neuroscience Education or communication techniques. No components of the "Algo(S)Therapy" program are included.
  Arms: Usual Physiotherapy Treatment

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of the "Algo(S)Therapy" Pain Neuroscience Education (PNE) program in patients with chronic musculoskeletal pain. The study will assess whether the integration of communication skills training for physiotherapists enhances the outcomes of PNE. Participants will be randomly assigned to one of three groups: (1) PNE with communication-focused delivery, (2) PNE without communication emphasis, or (3) standard- usual physiotherapy care. The primary objective is to determine whether PNE combined with enhanced communication skills leads to greater improvements in pain, function, and psychosocial outcomes compared to the other interventions.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of the "Algo(S)Therapy" Pain Neuroscience Education (PNE) program in the management of chronic musculoskeletal pain (CMP), with a focus on the added value of physiotherapists' communication skills. The study will be conducted in accordance with the CONSORT guidelines.

Eligible participants will be men and women aged 18 to 65 years, diagnosed with chronic musculoskeletal pain in the lumbar spine, neck, shoulder, or knee for more than 3 months, reporting a pain intensity ≥3/10 on the Numeric Pain Rating Scale (NPRS), and experiencing symptoms on most days of the week. All participants must be fluent in the Greek language. Exclusion criteria include acute pain, neurological or neuromuscular disorders, malignancy, recent surgeries or fractures within the past year, fibromyalgia, pregnancy, corticosteroid use, cognitive impairments that affect communication or questionnaire completion, or participation in other therapeutic programs during the study period.

Participants will be randomized into one of three groups:

Experimental Group 1: Participants will receive individualized PNE-based physiotherapy delivered by physiotherapists who have completed the full "Algo(S)Therapy" program, which includes both pain neuroscience and communication skills training specific to managing patients with chronic pain.

Experimental Group 2: Participants will receive the same PNE-based physiotherapy intervention, but from physiotherapists who have completed only the pain neuroscience component of the "Algo(S)Therapy" program. These therapists will not have received any training in communication skills or related modules.

Control Group will receive standard physiotherapy treatment without any exposure to PNE or communication-focused training.

All therapists in the experimental groups will have at least two year of experience treating patients with chronic musculoskeletal pain and will be selected based on performance in the "Algo(S)Therapy" training program. The intervention for all groups will last five weeks, with two sessions per week (total of 10 sessions).

The study will utilize validated outcome measures to evaluate pain, function, psychosocial variables, and therapeutic alliance. These include:

Numeric Pain Rating Scale (NPRS) Pain drawings (APDs) Central Sensitization Inventory (CSI) Pain Catastrophizing Scale (PCS) Tampa Scale for Kinesiophobia (TSK) Brief Illness Perception Questionnaire (B-IPQ) Pain Self-Efficacy Questionnaire (PSEQ) Pittsburgh Sleep Quality Index (PSQI) State-Trait Anxiety Inventory (STAI) Oswestry Disability Index (ODI) Working Alliance Inventory - Short Revised (WAI-SR) Satisfaction of treatment (Global Rating of Change - GroC) Days with disability (Recorded in an electronic data collection notebook) Adherence to Intervention (Recorded electronically) Adverse Effects (Recorded electronically)

Assessments will be conducted at three time points: baseline (pre-intervention), post-intervention, and 3-month follow-up. Statistical analysis will include repeated measures ANOVA to evaluate within- and between-group differences over time. The required sample size of 90 participants was calculated using G*Power, accounting for an estimated 10% dropout rate.

The main goal of this study is to determine whether the inclusion of communication training in a PNE-based physiotherapy program can significantly enhance clinical outcomes in patients with chronic musculoskeletal pain, compared to PNE alone or standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Diagnosis of chronic musculoskeletal pain in the lumbar spine, cervical spine, shoulder, or knee
* Pain duration longer than 3 months
* Pain intensity ≥3/10 on the Numeric Pain Rating Scale (NPRS)
* Pain present most days of the week
* Able to understand and speak the Greek language

Exclusion Criteria:

* Acute pain in any body region
* Neurological disorders or myopathies
* Chronic pain of non-musculoskeletal origin
* Active cancer diagnosis
* History of trauma, fractures, or surgery in the past year
* Pregnancy
* Diagnosis of fibromyalgia
* Cognitive impairments affecting communication or completion of questionnaires
* Current use of corticosteroid medication
* Participation in other treatment programs or alternative therapies during the study period
* Concurrent enrollment in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both men and women aged 18 to 65 years, who meet the inclusion criteria for chronic musculoskeletal pain, are eligible for participation in this study.
Enrollment: 90 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale - NPRS | Baseline, Post-intervention (Week 5), and 3-Month Follow-Up
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), where participants rate their average pain on a scale from 0 (no pain) to 10 (worst imaginable pain). The measure will be used to determine the effectiveness of each intervention in reducing chronic musculoskeletal pain.

SECONDARY OUTCOMES:
Central Sensitisation Inventory (CSI) | Baseline, Post-intervention (Week 5), and 3-Month Follow-Up
  The CSI assesses symptoms related to central sensitization in chronic pain conditions. The score ranges from 0 to 100, with higher scores indicating greater sensitization.
Pain Catastrophizing Scale (PCS) | Baseline, Post-intervention (Week 5), and 3-Month Follow-Up
  The PCS evaluates negative cognitive and emotional responses to pain, including rumination, magnification, and helplessness. Scores range from 0 to 52, with higher scores indicating greater levels of pain catastrophizing. This measure helps assess the psychological effect of the intervention.
Tampa Scale for Kinesiophobia (TSK) | Baseline, Post-intervention (Week 5), and 3-Month Follow-Up
  The TSK measures fear of movement or re-injury, which can limit function in individuals with chronic pain. Scores range from 17 to 68, with higher scores reflecting greater kinesiophobia. This outcome examines whether the intervention improves patients' movement confidence.
Pain Sensitivity Questionnaire (PSQ) | Baseline, Week 5, and 3-Month Follow-Up
  The PSQ assesses self-reported pain sensitivity through imagined everyday painful situations. It helps identify individuals with increased pain perception, a factor often present in chronic pain conditions. The total score ranges from 0 to 10, with higher scores indicating greater pain sensitivity. This outcome evaluates whether the intervention influences pain sensitivity levels.
Pain Self-Efficacy Questionnaire (PSEQ) | Baseline, Week 5, and 3-Month Follow-Up
  The PSEQ assesses a patient's confidence in performing activities despite their pain. Scores range from 0 to 60, with higher scores indicating stronger pain self-efficacy. This outcome evaluates the empowering effect of the intervention.
Brief Illness Perception Questionnaire (B-IPQ) | Baseline, Week 5, and 3-Month Follow-Up
  The B-IPQ measures patients' perceptions of their illness across cognitive and emotional dimensions. The total score ranges from 0 to 80, with higher scores indicating more negative or threatening views of their pain condition. This outcome assesses changes in illness perception related to the intervention.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 5, and 3-Month Follow-Up
  The PSQI evaluates sleep quality over the past month. It generates a global score ranging from 0 to 21, where scores above 5 indicate poor sleep quality. This outcome assesses whether the intervention contributes to improved sleep in chronic pain patients.
State-Trait Anxiety Inventory (STAI) | Baseline, Week 5, and 3-Month Follow-Up
  The STAI measures both current (state) and general (trait) anxiety. Each subscale yields a score from 20 to 80, with higher scores reflecting greater anxiety levels. This outcome helps evaluate the intervention's impact on anxiety associated with chronic pain.
Pain Disability Index (ODI) | Baseline, Week 5, and 3-Month Follow-Up
  Pain-related disability will be assessed using the Pain Disability Index (PDI), a 7-item questionnaire that evaluates interference from pain in major life domains. Each item is scored from 0 (no disability) to 10 (total disability), with a total score range of 0-70. Higher scores indicate greater functional impairment.
Working Alliance Inventory - Short Revised (WAI-SR) | Week 5 (Post-intervention only)
  The WAI-SR assesses the quality of the therapeutic alliance between the physiotherapist and the patient. Scores range from 12 to 84, with higher scores indicating a stronger working alliance. This measure is collected post-intervention to evaluate the interpersonal impact of the therapist's communication skills.
Satisfaction with Treatment (Global Rating of Change - GROC) | Post-intervention (Week 5) and 3-Month Follow-Up
  Participants will rate their perceived overall change in condition using the Global Rating of Change (GROC) scale, which typically ranges from -7 ("a very great deal worse") to +7 ("a very great deal better"). This outcome assesses overall patient satisfaction and perceived treatment effectiveness.
Pain Medication Consumption | Weekly during the 5-week intervention and at 3-Month Follow-Up
  Participants will report their use of pain medication throughout the intervention period. Data will be recorded electronically frequency. This outcome assesses whether the intervention reduces reliance on pharmacological pain management.
Adherence to Intervention | Throughout the 5-week intervention period
  Adherence will be tracked electronically by recording participant attendance to scheduled sessions. This outcome measures compliance with the intervention protocol.
Adverse Effects | Monitored continuously throughout the 5-week intervention
  Any adverse effects related to the intervention-such as increased pain, emotional distress, or any unexpected physical or psychological responses-will be reported by participants and recorded electronically. This outcome assesses the safety and tolerability of the interventions from a patient-reported perspective and supports real-time monitoring by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, Professor, Study Chair — Physiotherapy Department, University of Thessaly, Greece
Locations (1):
- Physiotherapy Department, University of Thessaly, Greece, Lamia, Central Greece, Greece